CLINICAL TRIAL: NCT07327697
Title: A Randomized, Double-blinded, Parallel, Positive-controlled Study to Compare the Pharmacokinetic, Safety and Immunogenicity of Single-dose QL2302 vs. Tezspire ® in Healthy Subjects
Brief Title: A Comparative Phase 1 Study to Evaluate the Pharmacokinetic and Safety of QL2302 vs. Tezspire® in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL2302-101
Record Dates: First submitted 2025-12-12; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
MeSH Terms: interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2302 (Experimental)
  Interventions: Drug: QL2302
- Tezspire® (Active Comparator)
  Interventions: Drug: Tezspire

INTERVENTIONS:
Drug: QL2302 — 210mg/1.91mL; single dose; subcutaneous injection
  Arms: QL2302
Drug: Tezspire — 210mg/1.91mL; single dose; subcutaneous injection
  Arms: Tezspire®

SUMMARY:
This is a randomized, double-blinded, controlled Phase 1 study to compare the pharmacokinetic, safety and immunogenicity of QL2302 versus Tezspire®（Tezepelumab） in healthy subjects after a single dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged from 18 to 45 years (including the boundary value), male and female.
2. Body weight 50.0-85.0 kg (including boundary value), and BMI 19.0-26.0 kg/m2 (including boundary value).
3. Normal results or abnormal results with no clinical significance of disease history/vital signs/laboratory examination/ECG according to the PI's judgment.
4. The subject (including partner) has no pregnancy plan or sperm donation plan during the whole trial period, and voluntarily adopts effective contraceptive measures.
5. Sign the informed consent before participating the study, and fully understand the content, process and possible risks.

Exclusion Criteria:

1. History of allergic reactions or hypersensitivity to Tezepelumab or excipients, or other biologics.
2. Donated at least 400 mL within 3 months prior to screening, or at least 200 mL within 4 weeks prior to the screening visit, or plan to donate blood during the study.
3. Smoked more than 5 cigarettes on average per day within 3 months prior to the screening visit.
4. Diagnosed as alcoholic, or subjects who consumed more than 14 units of alcohol per week within 6 months before the screening visit, or with positive alcohol test result on Day-1.
5. Drug abusers within 1 year prior to the screening visit, or subjects with positive urine drug test result during the screening period or on Day-1.
6. History of hospitalization due to infection or receiving anti-infection therapy through intravenous within 8 weeks prior to the screening visit, or had infection within 2 weeks prior to the screening visit.
7. Diagnosed a helminth parasitic infection within 6 months prior to the screening visit that has not been treated or has not responded to standard of care therapy.
8. History of active TB infection or a positive TB test result during screening period.
9. History of malignancy (except for NMSC treated with apparent success ≥5 years prior to screening).
10. Diagnosed with disease with abnormal clinical manifestations that should be excluded as judged by the PI.
11. History of treated by Tezepelumab or other TSLP-targeted biologics.
12. Have used prescription, OTC, herbal medicine, or health supplement within 2 weeks prior to randomization.
13. Vaccination with a live vaccine within 4 weeks or a attenuated vaccine within 2 weeks prior to randomization.
14. Have used biologics within 3 months prior to randomization, or within 5 half-life period before randomization. (whichever is longer)
15. Receiving treatment with any investigational product within 3 month prior to randomization or in 5 half-life period (whichever is longer), or treatment with any investigational equipment within 3 month prior to randomization.
16. Positive HbsAg, or HCV-Ab, or TPAb, or HIV antibody tests.
17. Female is pregnant or breastfeeding, or female who have not taken effective contraceptive measures within 14 days prior to randomization, or female with positive blood pregnant test.
18. Other conditions that considered inappropriate for participating the study, as per the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics Endpoint | Day 1-Day 134
  Peak plasma concentration (Cmax)
Pharmacokinetics Endpoint | Day 1-Day 134
  Area under the plasma concentration versus time curve from time 0 to infinity (AUC0-∞)